CLINICAL TRIAL: NCT06456398
Title: Advancing Interactive Medical Education of Anatomy Via the Metaverse Virtual 3D Printing Platform
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202402100RINE
Record Dates: First submitted 2024-05-28; First posted 2024-06-13 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-05

CONDITIONS: Virtual Reality
Keywords: Metaverse; Medical education; Anatomy; Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2D (traditional method) (No Intervention): Learning advanced anatomy using the traditional method of "using flat diagrams to correlate with computed tomography scans.
- 3D (Metaverse Virtual 3D Printing System) (Experimental): Learning advanced anatomy using the "Metaverse Virtual 3D Printing System" in virtual reality.
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — Through a randomized controlled trial, educational training will be designed, and pre- and post-tests will be conducted to compare the effectiveness of learning advanced anatomy using the "Metaverse Virtual 3D Printing System" in virtual reality, versus the traditional method of "using flat diagrams to correlate with computed tomography scans."
  Arms: 3D (Metaverse Virtual 3D Printing System)

SUMMARY:
The study aims to recruit 100 National Taiwan University 5th grade medical students who have completed a comprehensive basic anatomy course and are just entering surgical clinical rotations. Through a randomized controlled trial, educational training will be designed, and pre- and post-tests will be conducted to compare the effectiveness of learning advanced anatomy using the "Metaverse Virtual 3D Printing System" in virtual reality, versus the traditional method of "using flat diagrams to correlate with computed tomography scans." The study will assess the impact on learning outcomes, motivation, and learning experience in advanced anatomy education. We anticipate a well-structured learning model that bridges the gap between foundational and clinical medical courses.

DETAILED DESCRIPTION:
Anatomy is an important component of medical education, especially during surgical clinical rotations. It is crucial for students to be able to correlate the knowledge from flat anatomical diagrams to medical images and actual three-dimensional structures. However, for students with limited experience, transforming unfamiliar anatomical structures from 2D to 3D can be challenging. In recent years, numerous studies have pointed out the significant benefits of using three-dimensional anatomical models in anatomy education. Furthermore, interactive educational tools have shown even greater advantages.

The metaverse is a collective virtual shared space created by the integration of the internet and the physical world. It offers substantial assistance in virtual reality and interactive learning. While repeatedly using physical 3D printing for different body parts can enhance the understanding of three-dimensional structures, it is costly and time-consuming. Thus, through the collaborative effort of National Taiwan University Hospital department of surgery and Graduate institute of networking and multimedia, National Taiwan University, the "Metaverse Virtual 3D Printing System" has been developed to allow medical students to use wearable devices for immersive learning of detailed, interactive anatomy in a virtual platform.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old studying in the Department of Medicine at National Taiwan University
* Completed a full one-year anatomy lecture course and gross anatomy internship in the third year at the Department of Medicine, National Taiwan University.
* Students who have not yet received a complete clinical internship in thoracic surgery.
* Recruit willing subject medical students during their internship in thoracic surgery

Exclusion Criteria:

* Cybersickness
* Person who is sensitive to light stimulation

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire of Learning self-efficacy assessment | 1 year
  The results of questionnaires do not collect personal information. The values of the questionnaire scale do not indicate good or bad results.
Questionnaire of Motivated Strategies for Learning (MSLQ) | 1 year
  The results of questionnaires do not collect personal information. The values of the questionnaire scale do not indicate good or bad results.
Questionnaire of Technology Acceptance Model (TAM) | 1 year
  The results of questionnaires do not collect personal information. The values of the questionnaire scale do not indicate good or bad results.
Pre- and post-test learning tests | 1 year
  The results of tests will not affect academic performance.

CONTACTS AND LOCATIONS:
Overall Officials: Xu-Heng Chiang, MD, Principal Investigator — National Taiwan University Hospital